CLINICAL TRIAL: NCT01917786
Title: Effect of Dexmedetomidine on QT Interval in Pediatric Patients Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00171
Record Dates: First submitted 2013-06-25; First posted 2013-08-07 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Surgery
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dexmedetomidine patients: Surgical patients receiving dexmedetomidine.
  Interventions: Device: ECG
- Control patients: Surgical patients not receiving dexmedetomidine.
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG

SUMMARY:
Various medications used in anesthesia have been implicated in the prolongation of QT interval. Recently, there has been an increase in the use of dexmedetomidine in patients presenting for surgeries given its beneficial sedative, anxiolytic, and analgesic properties. It has several desirable properties including minimal respiratory side effects as well as the ability to decrease intraoperative and postoperative analgesic requirements. In many of the patients who present for routine surgical procedures, dexmedetomidine is a common component of their anesthetic care. This is a study to assess the effects of dexmedetomidine on the QT interval in children presenting for surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade 1 or 2.
* Scheduled to receive dexmedetomidine.

Exclusion Criteria:

* Known allergy to dexmedetomidine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving dexmedetomidine as part of their surgical anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in QT interval | Baseline, 5 mins., 10 mins.
  ECG will be done to assess QT interval prior to induction (baseline), after induction (5 mins.) and after dexmedetomidine (10 mins.)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Kako H, Krishna SG, Sebastian R, Smith K, Tobias JD. Effect of dexmedetomidine on the QT interval in pediatric patients undergoing general anesthesia. J Anesth. 2015 Dec;29(6):862-7. doi: 10.1007/s00540-015-2056-2. Epub 2015 Aug 4. PMID 26238761